CLINICAL TRIAL: NCT04180124
Title: Movement Analysis of Stroke Patients When Walking on a Treadmill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-1349
Record Dates: First submitted 2019-10-21; First posted 2019-11-27 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-01

CONDITIONS: Stroke
Keywords: Gait pattern; Treadmill walking; Arm swing
MeSH Terms: conditions — Stroke | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- GaitRite (Experimental): Patients will walk on the GaitRite.
  * forward walking at comfortable gait speed (6 x 10 meter)
  * backward walking at comfortable gait speed (4 x 10 meter)
  Interventions: Other: Walking
- Treadmill walking self-paced (Experimental): Patients will walk on the treadmill in self-paced mode. They can control walking speed by themselves.
  Patient walks for 3 minutes for every condition = data will be recorded for 1 minute.
  Interventions: Other: Walking
- Treadmill walking fixed speed - comfortable speed (Experimental): Patients will walk on the treadmill in fixed speed mode. They will walk at comfortable gait speed, which is determined in the familiarization period.
  Patient walks for 3 minutes for every condition = data will be recorded for 1 minute.
  Interventions: Other: Walking
- Treadmill walking fixed speed - fast speed (Experimental): Patients will walk on the treadmill in fixed speed mode. They will walk at a gait speed, which is 1 minimal clinical difference faster than their comfortable gait speed.
  Patient walks for 3 minutes for every condition = data will be recorded for 1 minute.
  Interventions: Other: Walking
- Treadmill walking fixed speed - backward walking (Experimental): Patients will walk on the treadmill in fixed speed mode. Patient will walk backwards on the treadmill if they are able to.
  Patient walks for 3 minutes for every condition = data will be recorded for 1 minute.
  Interventions: Other: Walking

INTERVENTIONS:
Other: Walking — Patients walk over ground on a mat with sensors and on a treadmill with sensors (in different conditions) to compare their movement pattern.
  Also the movement pattern will be compared between walking at comfortable walking speed en fast walking.
  Finally, the correlation between upper extremity impairment and arm swing will be investigated.

SUMMARY:
In daily clinic, the use of treadmills to analyze the gait quality of a patient increases. The advantages of using a treadmill are that a smaller space is needed compared to a 3D lab for motion analysis, more steps can be recorded in shorter time period and patients should not start, stop or rotate during the analyses. One of the systems which can be used to perform motion analysis on a treadmill is the GRAIL. This GRAIL (Gait Real-time Analysis Interactive Lab) consists of an advanced treadmill with force sensors. Patients can walk on this treadmill with an imposed speed (fixed-speed) or at a speed determined by the patient itself (self-paced). Because not everyone is used to walk on a treadmill it is important to know if a person's walking pattern is different when he walks over ground compared to walking on the treadmill. Based on these insights, decisions can be made regarding interventions including treadmill training or this findings can be taking into account during further analysis of walking patterns on a treadmill. For this study stroke patients would be invited for an assessment on the treadmill (1 assessment moment). The movement pattern of these patients would be compared in different conditions:

* (Forward and backward) Walking at comfortable walking speed on the GAITRite
* Walking at comfortable walking speed on the treadmill in fixed speed mode
* Walking at comfortable walking speed +0.2 m/s (faster walking) on the treadmill in fixed speed mode
* Walking at comfortable walking speed on the treadmill in self-paced mode
* Backward walking at comfortable walking speed on the treadmill in fixed speed mode (only if patients are eligible to do so)

Hypotheses based on this study protocol:

* Do stroke patients walk different over ground compared to treadmill walking
* Do stroke patients walk different during treadmill walking self-paced compared to fixed speed
* Do stroke patients walk different during treadmill walking fixed speed comfortable walking speed compared to fast walking
* Is there a correlation between upper extremity impairment and arm swing

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients with the ability to walk without walking devices for 6 minutes without rest (indoor walking). Use of AFO is allowed if necessary.

Exclusion Criteria:

* Traumatic brain lesions (car accident, fall with bike, …)
* Other disorders such as neurologic, musculoskeletal, respiratory or severe cardiovascular disorders that affected gait performance

  * Bilateral stroke
  * Cerebellar stroke
  * Orthopedic surgery lower limbs in the past
  * Cognitive or language impairments that prevent the patients from understand simple orders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Change in kinematics | Single point of assessment in one day
  Change in full body 3D kinematic analyses during walking (°)
Change in kinetics | Single point of assessment in one day
  Change in full body 3D kinetic analyses during walking

SECONDARY OUTCOMES:
Speed variability during self-paced treadmill walking | Single point of assessment in one day
  Average walking speed (and standard deviation) during self-paced treadmill walking
Postural stability test | Baseline assessment before walking trials
  Balance test
Fugl Meyer assessment UL | Baseline assessment before walking trials
  Impairment test for upper extremity in stroke patients: Fugl Meyer assessment - score between 0 and 66. Higher score reflects less impairment of the upper limb.
Fugl Meyer assessment LL | Baseline assessment before walking trials
  Impairment test for lower extremity in stroke patients: Fugl Meyer assessment lower extremity. Scores between 0 - 34. Higher score reflects less impairment of the lower limb.
Lateral rotation of the scapula | Baseline assessment before walking trials
  Lateral rotation of the scapula measured with an inclinometer (°)

OTHER OUTCOMES:
Demographic variables | Before walking trials
  gender, age, stroke type, stroke date, hemiparetic side, use of walking aids for outdoor walking

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No